CLINICAL TRIAL: NCT04901741
Title: An Open-label Phase 2 Study of Olaptesed Pegol (NOX-A12) Combined With Pembrolizumab and Nanoliposomal Irinotecan/5-FU/Leucovorin or Gemcitabine/Nab-paclitaxel in Microsatellite-stable Metastatic Pancreatic Cancer Patients
Brief Title: Olaptesed With Pembrolizumab and Nanoliposomal Irinotecan or Gemcitabine/Nab-Paclitaxel in MSS Pancreatic Cancer
Acronym: OPTIMUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNOXA12C701; 2021-001963-25 (EudraCT Number); KEYNOTE-B01 (Other: Merck Sharp & Dohme LLC); MK-3475-B01 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — NOX-A12; pembrolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: olaptesed pegol + pembrolizumab + nanoliposomal irinotecan + 5-FU + LV (Experimental)
  Interventions: Drug: Olaptesed pegol; Drug: Pembrolizumab
- Arm 2: olaptesed pegol + pembrolizumab + gemcitabine + nab-paclitaxel (Experimental)
  Interventions: Drug: Olaptesed pegol; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Olaptesed pegol — 400 mg per week as continous infusion until progression or intolerable toxicity
  Other Names: NOX-A12
Drug: Pembrolizumab — 200 mg every 3 weeks as i.v. infusion until progression or intolerable toxicity or a maximum of 35 administrations
  Other Names: KEYTRUDA®

SUMMARY:
The purpose of this study is to provide a go/no-go decision for a randomized expansion study by assessing the disease control rate (DCR) at 6 weeks for the combination of olaptesed pegol on top of pembrolizumab and (Arm 1) nanoliposomal irinotecan, 5-FU and leucovorin or (Arm 2) gemcitabine and nab-paclitaxel, to assess safety and tolerability and time-to-event endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed microsatellite-stable tumor pathology, if data available
* Patient with histologically or cytologically confirmed primary metastatic adenocarcinoma of the pancreas, who

  1. Arm 1: stopped first-line treatment with gemcitabine/nab-paclitaxel after documented objective radiographic progression OR
  2. Arm 2: stopped first-line treatment with FOLFIRINOX or modified FOLFIRINOX after documented objective radiographic progression
* Measurable disease based on RECIST 1.1 as determined by the investigational site
* Estimated minimum life expectancy 3 months
* Eastern Cooperative Oncology Group (ECOG) performance score 0 to 1
* Adequate organ function laboratory values within the ranges specified: Serum albumin ≥ 3.0 g/dL; Hematological system: Hemoglobin (Hb) ≥ 9.0 g/dL or ≥5.6 mmol/L, Absolute neutrophil count (ANC) ≥ 1,500/mm³, Platelets ≥ 100,000/mm³; Renal system: Creatinine ≤ 1.5 x ULN OR eGFR ≥30 mL/min for patient with creatinine levels >1.5 × institutional ULN; Hepatic system: Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN, ALT and AST ≤ 2.5 x ULN (≤5 × ULN for patients with liver metastases); Coagulation: INR OR PT ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants, aPTT ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter, prior to treatment.
* Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Patients with ≤ Grade 2 neuropathy may be eligible. Patients with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
* If the patient had major surgery, the patient must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention
* Prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and discontinued from that treatment due to a Grade 3 or higher irAE
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines are allowed
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or current pneumonitis / interstitial lung disease
* Active infection requiring systemic therapy
* Known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Previous allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Go/no-go decision for a randomized expansion study | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
  Assessment of the disease control rate (DCR) at 6 weeks for the combination of olaptesed pegol on top of pembrolizumab and (Arm 1) nanoliposomal irinotecan, 5-FU and leucovorin or (Arm 2) gemcitabine and nab-paclitaxel

SECONDARY OUTCOMES:
Safety and tolerability | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
  Safety and tolerability of olaptesed pegol pegol on top of pembrolizumab and (Arm 1) nanoliposomal irinotecan, 5-FU and leucovorin or (Arm 2) gemcitabine and nab-paclitaxel
DCR at 12 weeks | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
Progression free survival (PFS) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
Overall response rate (ORR) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
median Overall survival (mOS) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
Duration of response (DOR) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
Time-to-best overall response (TBOR) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab
Time-to-next-anticancer-treatment (TTNT) | until progression or intolerable toxicity to completion of 35 administrations (approximately 2 years) with pembrolizumab